CLINICAL TRIAL: NCT02108912
Title: The Impact of Gait Training on the Metabolic Costs of Walking and Cardiorespiratory Capacity in Persons Post Stroke
Brief Title: Metabolic Costs of Walking Post Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHA CV study; AHA Award #14CRP18500016 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2014-03-28; First posted 2014-04-09 (Estimated); Results first posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2018-10

CONDITIONS: Acute Stroke
Keywords: stroke; gait; cardiovascular
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional outpatient (Experimental): Traditional outpatient physical therapy
  Interventions: Other: Traditional outpatient
- ESTT outpatient (Experimental): ESTT (early standardized task-specific training) in outpatient rehabilitation
  Interventions: Other: ESTT

INTERVENTIONS:
Other: ESTT — ESTT is early-standardized task-specific training is a treadmill and over ground gait protocol for gait recovery after stroke
  Arms: ESTT outpatient
Other: Traditional outpatient — Traditional physical therapy includes standard of care for gait recovery after stroke such as pre-gait activities, standing balance activities, strengthening, walking with assistive devices.
  Arms: Traditional outpatient

SUMMARY:
This will be a randomized, matched-group study to compare the cardiopulmonary / metabolic benefits for persons post stroke that learn to walk utilizing early treadmill training post-acute stroke to persons post stroke that learn to walk utilizing non-treadmill based gait training during the same time period. Participants (n=30) will be adults who have completed acute rehabilitation following a stroke. Random assignment will be to either the ESTT or traditional gait training protocol during the outpatient rehabilitation phase.

1. Group A: Traditional outpatient therapy (n = 15)
2. Group B: Treadmill training (ESTT) outpatient therapy (n = 15)

DETAILED DESCRIPTION:
At the time of enrollment, participants will be randomly assigned to one of the two groups depending on the severity of impairment in the hemiparetic lower extremity. Groups will be matched based on high functioning vs. low functioning (STREAM scores). Group assignment will be done by random drawing from concealed envelopes with red or blue chips for assignment to ESTT or non-treadmill based outpatient therapy services. For the next participant who is screened with a similar STREAM impairment level, he/she will be placed in the alternate group to match the group assignments. Enrollment will proceed in this fashion. All outpatient therapy services will be provided at the UT Southwestern School of Health Professions School of Physical Therapy Gait Disorders Clinic (UTSW GDC). The groups will be as follows:

1. Group A: Traditional outpatient therapy (n = 15)
2. Group B: Treadmill (ESTT) outpatient therapy (n = 15) Therapy for the purposes of the study will be discontinued after a maximum of 24 training sessions or 8 weeks. It is anticipated, based on the research concerning AFO use in persons with stroke, that all participants will require an AFO for safe gait training in the outpatient setting.

Traditional outpatient therapy: For persons in Group A, gait training will consist of 30 minutes of walking training. The program may include a variety of interventions that are commonly done to rehabilitate gait after stroke (excluding treadmill training). Walking may include the use of various assistive devices such as rolling walkers, gait trainers, canes and crutches. Other tools that may be utilized include visual cues (tape, lasers) and auditory cues (metronome). Other activities such as single limb stance and stair climbing may be included to facilitate limb stability. Functional electrical stimulation (FES) may be used to facilitate muscle activation in the hemiparetic lower extremity during gait training for all participants. Stimulation may be applied to muscles of the upper and/or lower leg gait training. Use of electrical stimulation will be documented, including all parameters (make and model of unit, rate of stimulation [pulses per second], waveform, and duration of use). Appropriate exercises from a bank of exercises will be selected for each participant. The bank of exercises will include: standing heel cord stretches, single leg stance, sit to stand, timed standing, marching in place, tap ups, step ups, step throughs, standing ball roll, stair climbing, standing Theraband exercises, wall squats. They will be advised to complete the exercises daily (5 days/week total) for a total of 30 minutes per day. In addition, they will be instructed to wear the AFO for all upright mobility tasks, in combination with the prescribed assistive device.

Treadmill (ESTT) outpatient therapy: For persons in Group B, study-related outpatient gait training will be initiated on the treadmill with partial body weight support. The initial body weight support will be set between 30% and 50% of patient's body weight. During progressive training sessions, the amount of body weight support will attempt to be reduced and the researcher will assess the response to the increased body weight on the gait pattern. The initial speed of the treadmill will be 0.7 mph (minimum initial speed) and will be increased progressively as tolerated until a speed of 1.8 mph is reached. Subject tolerance to the intervention will be monitored closely. Gait training on the treadmill will be scheduled in 30-minute sessions. The subjects will be allowed to take rest breaks as needed during the treadmill training.

During gait training on the treadmill, ankle control will be facilitated by means of an ankle foot orthosis (AFO) with a double adjustable joint. For over ground gait, participants will also use an AFO with a double adjustable joint Functional electrical stimulation (FES) may be used to facilitate muscle activation in the hemiparetic lower extremity during gait training for all participants. Over ground gait will not be initiated until the subject is able to walk on the treadmill with no more than 10% body weight support and with no more than minimal assist to advance the hemiparetic leg at a speed of 0.8 mph or greater for at least 3 minutes for two consecutive bouts. (Subjects can also have assistance with weight shift.) Once over ground gait is initiated, either bilateral or unilateral support will be used, depending on upper extremity control and general upright stability. If the quality of the gait deteriorates significantly from the gait observed on the treadmill, over ground gait will be halted for that session. Treadmill training will continue to progress to over ground gait. Once over ground gait training is initiated, 20 minutes of the 30 total therapy minutes will be spent on treadmill training and 10 minutes will be spent on over ground gait training. Treadmill training will continue until subjects are able to walk 10 minutes without resting with no body weight support, but with vest on for safety, without upper extremity support without assist for weight shift or lower extremity control at a speed of 1.8 mph. If this is prior to the conclusion of study-related therapy, the entire 30 minute session will be spent practicing over ground gait.

Appropriate exercises from a bank of exercises will be selected for each participant. The bank of exercises will include: standing heel cord stretches, single leg stance, sit to stand, timed standing, marching in place, tap ups, step ups, step throughs, standing ball roll, stair climbing, standing Theraband exercises, wall squats. They will be advised to complete the exercises daily (5 days/week total) for a total of 30 minutes per day. In addition, they will be instructed to wear the AFO for all upright mobility tasks, in combination with the prescribed assistive device.

The Step Program: To introduce this component of the study, the participant and caregiver/support person will be given a 15-minute presentation entitled Step it Up. This program was developed by the research team and it addresses the critical need and benefits of exercise for persons post stroke, methods of safe exercise monitoring and information on progression of exercise intensity and duration to improve cardiorespiratory function. The presentation will include an explanation of the Borg Rate of Perceived Exertion (RPE, 6-20 scale) and directions on how to utilize a pedometer for daily walking measurement. Following the presentation, participants will meet with an investigator and demonstrate competency with the application of the pedometer and utilization of the RPE scale. Each participant will be provided written material that covers the salient points of the presentation. They will also receive a notebook that has the instructions along with 16 weekly logs for recording walking data. The training should take approximately 30 minutes and will take place following the final gait treatment.

The walking program will continue until T4 and T4a. Each participant will be scheduled for this testing within 10 calendar days of the 24-week anniversary of the commencement of outpatient therapy. At this testing time (T4 & T4a) all outcome measures will be repeated. The final testing time (T5 and T5 a) will be completed within 10 calendar days of 288-day anniversary of commencement of outpatient physical therapy. All outcome measures will be repeated at this testing time. This will be the termination point of the study.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of recent cerebrovascular accident (CVA) (less than 6 weeks post at the time of admission to inpatient rehabilitation)
* able to give informed consent independently or have family member or other authorized surrogate available to give consent
* first time stroke OR complete gait recovery from prior stroke
* sufficient support at home to participate in home-based fitness training program
* transportation to University of Texas Southwestern Medical Center Gait Disorders Clinic (UTSW GDC) for therapy and testing
* ability to follow one-part commands

Exclusion Criteria:

* non-ambulatory before onset of stroke (at time of admission to inpatient rehabilitation)
* bilateral stroke
* presence of severe cardiac problems (heart failure [New York Heart Association > Class 2], unstable or exercise-induced angina)
* other co-morbidities which could affect gait training (i.e. amputation, spinal cord injury, traumatic brain injury, etc.)
* recent myocardial infarct (within 4 weeks of date of inpatient rehabilitation admission)
* any uncontrolled health condition for which exercise is contraindicated
* severe lower extremity joint disease/pathology that would interfere with gait training
* subjects -with body mass index (BMI) greater than 40
* significant cognitive impairment (less than 2 on the Functional Independence Measure [FIM] cognitive sub-scale)
* age greater than 80 years or less than 18 years
* able to complete 5 or more full heel raises with the affected ankle in standing with the knee extended with no more than one or two fingers on support surface for balance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen J McCain, DPT, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern School of Health Professions, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Traditional Outpatient | ESTT Outpatient
Started | 9 | 7
Completed | 6 | 6
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — lack of transportation | 1 | 0
Not completed — high blood pressure | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional Outpatient | ESTT Outpatient | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Continuous [Mean (Full Range); unit: Years] | 53.7 [42 to 65] | 53.4 [38 to 68] | 53.6 [38 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Maximum Exercise Tolerance Testing
Description: Exercise tests will be performed with a treadmill with a static/dynamic body weight system. Measurements will be conducted with open circuit spirometry. Heart rate will be continuously monitored by electrocardiogram. Blood pressure will be monitored every 2 minutes. Participants will be allowed a 3-minute warm-up. Following the warm-up, participants will be allowed up to 10 minutes to rest or until they recovery to baseline heart rate, respiration rate and blood pressure.
Time Frame: Change in exercise tolerance from enrollment to 9 weeks later and 25 weeks later
Population: The data was corrupted and unable to be analyzed.
Arm/Group | Traditional Outpatient | ESTT Outpatient
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in 6-Minute Walk Test Distance
Description: Each subject will be asked to complete a 6-Minute Walk test. They will be advised to walk at a pace they think they can maintain for the entire time. Resting is permitted provided they are not required to sit. Participants will not be given any verbal encouragement during the test. A stop watch will be used to time the test and the distance will be measured with a calibrated measuring wheel along a 150 foot corridor. Heart rate will be monitored during the test by means of a Polar chest strap and values will be recorded at each minute of the test. Perceived rate of exertion using the Borg scale of 6-20 will be recorded at rest and each minute of the test.34 Blood pressure using an automated arm cuff will be recorded before and after the test.
Time Frame: At enrollment and week 25.
Population: The Borg and blood pressure measures were used to monitor the response of the participants to the activity. If the blood pressure rose too high, for example, testing was terminated. Likewise, if the Borg rating was too high, participants were allowed to rest and vital signs were assessed again.
Measure: Mean (Full Range); unit: feet
Arm/Group | Traditional Outpatient | ESTT Outpatient
Number analyzed (Participants) | 6 | 6
feet | 469.3 [128 to 661] | 529.2 [160 to 969]

3. Other Pre Specified Outcome: Temporal Spatial Gait Analysis
Description: Testing will be completed using a 14'x4', 16-level pressure sensing Zeno Walkway. This system utilizes a computerized gait system for data collection. Gait parameters that will be collected include center of pressure, center of mass, step/stride length, velocity, toe in/out, cadence, and left/right lower extremity ratios. Participants will be asked to walk at self-selected and safe fast walking paces for repeated straight direction walking trials to collect an average of 100 feet of straight distance. This testing will be done at T1, T2, T3 and T4. This test takes 15 minutes to complete.
Time Frame: At enrollment, week 9, week 17 and week 25.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Data was collected for a period of 2.5 years
Arm/Group | Traditional Outpatient | ESTT Outpatient
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 0/9 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No